CLINICAL TRIAL: NCT00954408
Title: Fatigue in Dystonia (IRB No. 108-2008)
Brief Title: Fatigue in Dystonia (a Single Session, Questionnaire-based Study of Fatigue in Dystonia)
Acronym: FID
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 108-2008
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Dystonia
MeSH Terms: conditions — Dystonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with dystonia: Patients with dystonia, 21-100 years of age.

SUMMARY:
The purpose of this study is to determine how common fatigue and sleepiness are in patients with dystonia.

DETAILED DESCRIPTION:
The purpose of the study is to determine the prevalence of fatigue in patients with dystonia. There are many factors which may impact fatigue but perhaps the most important of these is sleep. It is therefore critical that we collect data on sleep habits and sleepiness to help interpret our data on fatigue. We will be using the Epworth Sleepiness Scale to assess daytime somnolence and the Parkinson's Disease Sleep Scale to assess the presence or absence of common sleep disorders affecting patients with movement disorders along with the Multidimensional Fatigue Inventory and the Fatigue Severity Scale.

ELIGIBILITY:
Inclusion Criteria: diagnosis of dystonia

* Informed consent to be contacted about research

Exclusion Criteria:

* None

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Current dystonia patients in our clinic between the ages of 21 and 100.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2009-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To determine the prevalence of fatigue and sleepiness in patients with dystonia. | At the time of their visit.

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Okun, M.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida Movement Disorders Center, Gainesville, Florida, United States